CLINICAL TRIAL: NCT07265011
Title: Prospective Validation of an AI-Driven Ultrasound-Based Method for Estimating Hepatic Steatosis Using MRI-Derived Fat Fraction as Reference in Pediatric Metabolic Dysfunction-Associated Steatotic Liver Disease
Brief Title: Ultrasound-Based Estimation of Hepatic Steatosis in Pediatric MASLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jae Won Choi (Other)
Responsible Party: Sponsor-Investigator, Jae Won Choi, Clinical Assistant Professor, Seoul National University Hospital
Organization: Seoul National University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SNUH-2312-148-1496
Record Dates: First submitted 2025-11-23; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: MASLD; Pediatric
Keywords: MASLD; NAFLD; Fatty Liver; Pediatrics
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver | interventions — Ultrasonography; Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Liver Ultrasound and MRI (Experimental)
  Interventions: Diagnostic Test: Ultrasound and MRI

INTERVENTIONS:
Diagnostic Test: Ultrasound and MRI — Participants undergo same-day liver imaging including conventional B-mode ultrasound, quantitative ultrasound, and magnetic resonance imaging (MRI).
  Conventional Ultrasound: B-mode imaging performed on three ultrasound systems (Canon Aplio i800, Philips EPIQ, and Supersonic AIXPLORER) to acquire grayscale liver images for artificial intelligence (AI) analysis.
  Quantitative Ultrasound: Attenuation imaging (ATI) and shear wave elastography/dispersion measurements performed to assess hepatic fat and stiffness.
  MRI: Proton density fat fraction (PDFF) measurement used as the reference standard for hepatic steatosis quantification.
  All imaging is performed on the same day for each participant to ensure temporal consistency across modalities and vendors.

SUMMARY:
The purpose of this study is to validate an artificial intelligence (AI)-based algorithm that estimates hepatic steatosis using ultrasound (US) B-mode images in pediatric participants with metabolic dysfunction-associated steatotic liver disease (MASLD). The MRI proton density fat fraction (MRI-PDFF) serves as the reference standard for hepatic fat quantification.

ELIGIBILITY:
Inclusion Criteria:

* participants aged 8 to 18 years clinically indicated for liver ultrasound examination to evaluate hepatic steatosis
* participants with suspected or known metabolic dysfunction-associated steatotic liver disease (MASLD)
* able to understand the study purpose and provide written informed consent (from both participant and legal guardian).
* agree to undergo same-day liver MRI examination in addition to the ultrasound

Exclusion Criteria:

* unable to cooperate with imaging procedures
* parent or legal guardian unable to understand the study explanation
* contraindications to MRI
* determined by the investigator to be otherwise unsuitable for participation after consultation

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2024-12-31 (Actual); Primary Completion 2025-09-23 (Actual); Study Completion 2025-09-23 (Actual)

PRIMARY OUTCOMES:
Agreement Between AI-Predicted Ultrasound Fat Fraction (AI-USFF) and MRI Proton Density Fat Fraction (MRI-PDFF) | At time of imaging (single visit)
  Reference standard: MRI-PDFF (percentage)
  - intraclass correlation coefficient (ICC)

SECONDARY OUTCOMES:
Correlation Between AI-USFF and MRI-PDFF | At time of imaging (single visit)
  Reference standard: MRI-PDFF (percentage)
  - Pearson correlation coefficient (r)
Diagnostic Performance of AI-USFF for MRI-Based Hepatic Steatosis Grades | At time of imaging (single visit)
  The diagnostic performance of AI-USFF for detecting mild, moderate, and severe hepatic steatosis, as defined by MRI-PDFF thresholds, will be evaluated using area under the receiver operating characteristic curve (AUC).
Inter-Vendor Reproducibility of AI-USFF | At time of imaging (single visit)
  Reproducibility of AI-USFF across the three ultrasound systems are assessed using the intraclass correlation coefficient (ICC [2,k]).

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea